CLINICAL TRIAL: NCT05491733
Title: A 3-Treatment, 3-Period, 6-Sequence Randomized Crossover Single-Dose Study Evaluating the Bioequivalence of High-Load and Low-Load Oral Tablet Formulations of Apx001 and the Effect of Food on the Absorption of Apx001 From the High-Load Tablet In Healthy Subjects
Brief Title: A Bioequivalence Study of APX001 High-load and Low-load Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: APX001-108; C4791008 (Other: Alias Study Number)
Expanded Access: NCT06433128 (Available)
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Invasive Fungal Infections
Keywords: fosmanogepix; candida; aspergillus; scedosporium; fusarium; mucorales; rhizopus
MeSH Terms: conditions — Invasive Fungal Infections; Torulopsis | interventions — APX001A

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- APX001 Treatment A (Active Comparator): Oral tablet with a 25% drug load (low-load) in fasted participants
  Interventions: Drug: APX001; Drug: APX001A
- APX001A Treatment B (Experimental): Oral tablet with a high drug load in fasted participants
  Interventions: Drug: APX001; Drug: APX001A
- APX001A Treatment C (Experimental): Oral tablet with a high drug load in participants that are not fasted.
  Interventions: Drug: APX001; Drug: APX001A

INTERVENTIONS:
Drug: APX001 — Low-load oral tablet
  Other Names: fosmanogepix
Drug: APX001A — High-load oral tablet
  Other Names: fosmanogepix

SUMMARY:
A study to learn about the bioequivalence (the biochemical similarity of two medicines that share the same active ingredient and desired outcome for patients) of the study medicine called APX001 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.0 and 32.0 kg/m2, inclusive.
* Minimum body weight of 50 kg.
* Screening hematology, clinical chemistry, coagulation, and urinalysis consistent with overall good health and having an estimated glomerular filtration rate (eGFR) >80 mL/min, based on creatinine clearance calculation by the Cockcroft-Gault formula.

Exclusion Criteria:

* Having any uncontrolled or active major systemic disease including, but not limited to: cardiovascular, pulmonary, gastrointestinal, metabolic, urogenital, neurological, immunological, psychiatric, or neoplastic disorder with metastatic potential.
* History or presence of neurological disorders including abnormal movements or seizures.
* History or presence of malignancy within the past year. Subjects who have been successfully treated with no recurrence of basal cell carcinoma of the skin or carcinoma in-situ of the cervix may be enrolled.
* Significant and/or acute illness or chronic infection, as judged by the investigator, including, but not limited to: upper airway infection, urinary tract infection, or skin infection within 30 days prior to the first study drug administration.
* Taking any drug or herbal CYP3A modulator (e.g., erythromycin; St. John's Wort) within 4 weeks (or 5 half-lives, whichever is longer) or any other nutrients known to modulate CYP3A activity (e.g., grapefruit juice; Seville orange) within 2 weeks prior to the first admission.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Predose, 0.5, 1, 2, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 36, 48, 168, and 312 hours post dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Predose, 0.5, 1, 2, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 36, 48, 168, and 312 hours post dose
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | Predose, 0.5, 1, 2, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 36, 48, 168, and 312 hours post dose
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] | Predose, 0.5, 1, 2, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 36, 48, 168, and 312 hours post dose
Area Under the Curve From Time Zero to 24 hours (AUC0-24) | Predose, 0.5, 1, 2, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 36, 48, 168, and 312 hours post dose
Percentage of Area Under the Curve Extrapolated to Infinity (%AUCextra) | Predose, 0.5, 1, 2, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 36, 48, 168, and 312 hours post dose
Plasma Decay Half-Life (t1/2) | Predose, 0.5, 1, 2, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 36, 48, 168, and 312 hours post dose
Apparent Terminal Elimination Rate Constant (λz) | Predose, 0.5, 1, 2, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 36, 48, 168, and 312 hours post dose
Apparent Total clearance, Calculated as Dose/AUCinf (CL/F) | Predose, 0.5, 1, 2, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 36, 48, 168, and 312 hours post dose
Apparent Volume of Distribution at Terminal Phase (Vz/F) | Predose, 0.5, 1, 2, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 36, 48, 168, and 312 hours post dose
Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Baseline through Day 14
Number of Participants With Change From Baseline in Laboratory Tests Results | Baseline through Day 14
Number of Participants With Clinically Significant Change in Vital Signs | Baseline through Day 14
Number of Participants With Clinically Significant Findings in Electrocardiogram (ECG) Abnormalities | Baseline through Day 14
Number of Participants With Abnormalities in Physical Examinations | Baseline through Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Marc Engelhardt, Study Director — Basilea Pharmaceutica International Ltd, Allschwil
Locations (1):
- Pharmaceuticals Research Associates, Inc, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No